CLINICAL TRIAL: NCT00594165
Title: An Open-Label Extension to the Double-Blind SP512 Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Subjects With Early-Stage Idiopathic Parkinson's Disease.
Brief Title: An Open-Label Extension Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Early-Stage Parkinson's Disease.
Acronym: SP512OL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0702; SP512OL
Record Dates: First submitted 2007-12-24; First posted 2008-01-15 (Estimated); Results first posted 2010-02-25 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2010-09

CONDITIONS: Early-Stage Parkinson's Disease
Keywords: Rotigotine
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): Rotigotine
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine trans-dermal patches:
  10 cm2 (2 mg/24 hours); 20 cm2 (4 mg/24 hours); 30 cm2 (6 mg/24 hours); 40 cm2 (8 mg/24 hours)
  Optimal dosing:
  During the first year:
  The maximum Rotigotine dose allowed is 6 mg/24 hours.
  After the first year: allowed dose increase of Rotigotine up to a maximum of 16 mg/24 hours.
  Other Names: Neupro

SUMMARY:
The objective of this open-label extension is to assess the safety and tolerability of long-term treatment of the rotigotine patch in subjects with early-stage idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
This is the open-label extension to the randomized, double-blind, placebo-controlled SP512 trial that assessed the efficacy and safety and tolerability of the Rotigotine patch in subjects with early-stage idiopathic Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed six months of maintenance treatment in the SP512 double-blind trial

Exclusion Criteria:

* Subjects who had an ongoing serious adverse event from SP512 double-blind trial that was assessed as related to study medication

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2002-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (42):
- United States (37):
  - Peoria, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Fountain Valley, California
  - Fresno, California
  - Los Angeles, California
  - Englewood, Colorado
  - Danbury, Connecticut
  - New Haven, Connecticut
  - Miami, Florida
  - Pompano Beach, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Henderson, Nevada
  - New Brunswick, New Jersey
  - Albany, New York
  - Louisville, New York
  - New York, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Upland, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Roanoke, Virginia
  - Milwaukee, Wisconsin
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vernon, British Columbia
  - Ottawa, Ontario
  - Saskatoon, Saskatchewan

REFERENCES:
- [Result] Elmer LW, Surmann E, Boroojerdi B, Jankovic J. Long-term safety and tolerability of rotigotine transdermal system in patients with early-stage idiopathic Parkinson's disease: a prospective, open-label extension study. Parkinsonism Relat Disord. 2012 Jun;18(5):488-93. doi: 10.1016/j.parkreldis.2012.01.008. Epub 2012 Feb 10. PMID 22326237
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An Open-Label Extension to Assess the Safety of Long-Term Treatment of Rotigotine in Subjects with Early-Stage Idiopathic Parkinson's Disease from June 2002 to November 2008
Pre-assignment Details: Subject 10806 received SP512OL study medication at the final visit of SP512DB but never returned to the clinic; this subject is excluded from the Safety Set.
Groups:
- Rotigotine: Optimal dosing for Rotigotine transdermal patches, once daily: Year 1, the maximum dose allowed is 6 mg/24 hours. After Year 1, a dose increase is allowed up to a maximum of 16 mg/24 hours.
Period: Overall Study
Arm/Group | Rotigotine
Started | 217
Completed | 0 (Study fully recruited. Completed upon market authorization and commercial availability of Neupro.)
Not Completed | 217
Not completed — Major protocol violation | 1
Not completed — Lack of Efficacy | 12
Not completed — Adverse Event | 52
Not completed — Unsatisfactory compliance of subject | 6
Not completed — Subject withdrew consent | 27
Not completed — Study ended per sponsor | 102
Not completed — Lost to Follow-up | 4
Not completed — Other: PI discretion | 5
Not completed — Other: Subject moving | 3
Not completed — Other: Brain surgery controlled symptoms | 1
Not completed — Other: House bound; can't get to clinic | 1
Not completed — Other: Subject enrolled in other trial | 1
Not completed — Other: Site terminated participation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rotigotine
Number analyzed (Participants) | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 119
  >=65 years | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 147
Region of Enrollment [Number; unit: participants]
  United States | 186
  Canada | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event During This Open-label Extension Study
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: 7 years
Population: Of the 217 subjects who entered the study, 216 are included in this summary based on the Safety Set (SS). Subject 10806 received SP512OL study medication at the final visit of SP512DB but never returned to the clinic; this subject is excluded from the Safety Set.
Measure: Number; unit: Subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 216
Subjects | 214

2. Secondary Outcome: Number of Subjects Who Withdrew From the Trial Due to an Adverse Event.
Description: as for outcome 1
Time Frame: 7 years
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 216
subjects | 52

3. Secondary Outcome: Mean Epworth Sleepiness Scale Score During the Open-label Extension.
Description: The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. The total ESS score is the sum of 8 item-scores and can range between 0 and 24. The higher the score, the higher the person's level of daytime sleepiness.
Time Frame: Visit 9 (end of year 1), Visit 13 (end of year 2), Visit 17 (end of year 3), Visit 21(end of year 4), Visit 25 (end of year 5), Visit 29 (end of year 6), End of Treatment (last study visit or early withdrawal visit)
Population: Of the 217 subjects who entered the study, 216 are included in this summary based on the Safety Set (SS). Subject 10806 received SP512OL study medication at the final visit of SP512DB but never returned to the clinic; this subject is excluded from the Safety Set. Last observation carried forward (LOCF) was utilized.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 216
Score on a scale
  Visit 9 (end of year 1) (n=209) | 7.3 (4.4)
  Visit 13 (end of year 2) (n=209) | 7.9 (4.9)
  Visit 17 (end of year 3) (n=209) | 8.2 (5.2)
  Visit 21 (end of year 4) (n=209) | 8.4 (5.0)
  Visit 25 (end of year 5) (n=209) | 8.8 (5.0)
  Visit 29 (end of year 6) (n=209) | 8.5 (5.0)
  End of Treatment (n=216) | 9.0 (5.4)

ADVERSE EVENTS:
Time Frame: Up to 7 years
Description: Subject 10806 received SP512OL study medication at the final visit of SP512DB but never returned to the clinic; this subject is excluded from the Safety Set. Adverse event terms may appear in both summaries given that the same adverse event term may be reported for different subjects as either serious or non-serious.
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 102/216
Other Adverse Events (participants affected / at risk) | 206/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=216)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Myocardial infarction (Cardiac disorders) | 6 (6)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Atrioventricular block third degree (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2)
Lower gastrointestinal haemmorrhage (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 6 (7)
Asthenia (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Application site reaction (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 5 (8)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Infection (Infections and infestations) | 2 (3)
Localised infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 5 (6)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (3)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Strernal fracture (Injury, poisoning and procedural complications) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram ST-T change (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (7)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parkinson's disease (Nervous system disorders) | 5 (7)
Parkinsonism (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 4 (5)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Carotid artery occulusion (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 3 (3)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Sleep attacks (Psychiatric disorders) | 2 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Accute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Obstructuve airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 2 (2)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=216)
Anaemia (Blood and lymphatic system disorders) | 17 (19)
Cataract (Eye disorders) | 25 (39)
Nausea (Gastrointestinal disorders) | 66 (110)
Vomiting (Gastrointestinal disorders) | 26 (44)
Constipation (Gastrointestinal disorders) | 37 (42)
Dyspepsia (Gastrointestinal disorders) | 19 (19)
Diarrhoea (Gastrointestinal disorders) | 17 (21)
Dry mouth (Gastrointestinal disorders) | 15 (16)
Oedema peripheral (General disorders) | 79 (121)
Application site erythema (General disorders) | 31 (34)
Application site pruritus (General disorders) | 19 (25)
Application site irritation (General disorders) | 14 (14)
Fatigue (General disorders) | 24 (27)
Upper respiratory tract infection (Infections and infestations) | 33 (49)
Nasopharyngitis (Infections and infestations) | 25 (30)
Sinusitis (Infections and infestations) | 17 (21)
Urinary tract infection (Infections and infestations) | 33 (56)
Influenza (Infections and infestations) | 17 (18)
Fall (Injury, poisoning and procedural complications) | 69 (142)
Excoriation (Injury, poisoning and procedural complications) | 12 (14)
Contusion (Injury, poisoning and procedural complications) | 15 (18)
Skin laceration (Injury, poisoning and procedural complications) | 15 (20)
Procedural pain (Injury, poisoning and procedural complications) | 14 (16)
Weight decreased (Investigations) | 14 (16)
Blood cholesterol increased (Investigations) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 53 (69)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 40 (63)
Neck pain (Musculoskeletal and connective tissue disorders) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 51 (82)
Joint swelling (Musculoskeletal and connective tissue disorders) | 15 (16)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 (25)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 (16)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 (12)
Somnolence (Nervous system disorders) | 116 (198)
Dizziness (Nervous system disorders) | 58 (80)
Paraesthesia (Nervous system disorders) | 16 (23)
Hypoaesthesia (Nervous system disorders) | 14 (21)
Headache (Nervous system disorders) | 21 (32)
Tremor (Nervous system disorders) | 19 (22)
Memory impairment (Nervous system disorders) | 14 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (17)
Balance disorder (Nervous system disorders) | 14 (16)
Dyskinesia (Nervous system disorders) | 12 (13)
Parkinson's disease (Nervous system disorders) | 12 (12)
Insomnia (Psychiatric disorders) | 47 (55)
Depression (Psychiatric disorders) | 38 (45)
Anxiety (Psychiatric disorders) | 24 (28)
Hallucination (Psychiatric disorders) | 20 (28)
Confusional state (Psychiatric disorders) | 17 (19)
Sleep disorder (Psychiatric disorders) | 14 (16)
Abnormal dreams (Psychiatric disorders) | 13 (16)
Obsessive-compulsive disorder (Psychiatric disorders) | 12 (14)
Micturition urgency (Renal and urinary disorders) | 14 (14)
Urinary incontinence (Renal and urinary disorders) | 12 (14)
Erectile dysfunction (Reproductive system and breast disorders) | 19 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (15)
Rash (Skin and subcutaneous tissue disorders) | 15 (17)
Hypertension (Vascular disorders) | 27 (27)
Orthostatic hypotension (Vascular disorders) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.